CLINICAL TRIAL: NCT06426134
Title: Pilot Study on Ketosis Impact on Signs and Symptoms of Schizophrenia and Bipolar Disorders
Brief Title: Ketosis Impact on Signs & Symptoms of Schizophrenia and Bipolar disorderS
Acronym: KISSeS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Collaborators: Parnassia Groep (Other); The University of Texas at Dallas (Other); University of Alberta (Other); EnLiSense (Unknown)
Responsible Party: Principal Investigator, Karin Huizer, Principal Investigator; MD, PhD, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: NL83836.018.23; 2024.0100 (Other: METC AUMC)
Record Dates: First submitted 2024-05-08; First posted 2024-05-23 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Schizophrenia and Related Disorders; Psychosis; Bipolar and Related Disorders; Manic Episode; Depressive Episode
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders; Bipolar and Related Disorders; Mania | interventions — (R)-3-hydroxybutyl (R)-3-hydroxybutyrate; maltodextrin; Fructose; Pectins; Alginates; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- dGK (Experimental): 1x50 g dGK ketone drink
  Interventions: Dietary Supplement: (R)-3-hydroxybutyl (R)-3-hydroxybutyrate)
- isocaloric carb control (Active Comparator): 1x isocaloric carbohydrate control drink
  Interventions: Other: Maltodextrin, Fructose, Pectin, Sodium alginate, Sodium chloride

INTERVENTIONS:
Dietary Supplement: (R)-3-hydroxybutyl (R)-3-hydroxybutyrate) — 1x50g ingestion of pure dGK
  Other Names: delta G Ketones (dGK)
  Arms: dGK
Other: Maltodextrin, Fructose, Pectin, Sodium alginate, Sodium chloride — Isocaloric carbohydrate control (active control)
  Other Names: Maurten Drink Mix 160
  Arms: isocaloric carb control

SUMMARY:
The goal of this clinical trial is to learn if a ketone drink can improve signs and symptoms of patients with a schizophrenia-spectrum disorder (SSD), or a bipolar-spectrum disorder (BD).

The main questions it aims to answer are:

Does a ketone drink improve information processing in patients with SSD/BD?

Other questions it aims to answer are:

Does a ketone drink improve cognitive functioning in patients with SSD/BD? Does a ketone drink improve metabolism and inflammation in patients with SSD/BD? Does a ketone drink affect circadian rhythm in patients with SSD/BD?

Research will compare the effects of the ketone drink with that of an isocaloric carbohydrate drink in the same patients ('cross-over').

Participants will:

1. drink a ketone drink and (after a wash-out period) an isocaloric control drink (randomized order); after each drink:

   * EEG/EMG to determine information-processing parameters (PPI and P300)
   * cognitive tests
   * visual analog scale of mood, energy levels, ability to focus
   * indirect calorimetry to determine use of energy substrate
   * blood draws
2. for 5 consecutive days:

   * wear a continuous glucose monitor (CGM)
   * wear a non-invasive passive sweat biomarker sensor (EnLiSense device)
   * register a diet and nicotine diary
   * saliva sampling (max. 5x/day)

ELIGIBILITY:
Inclusion Criteria:

* Patients with a first-episode psychosis (underlying schizophrenia-spectrum disorder), or patients with a (hypo)manic or depressive episode (underlying bipolar disorder)
* Age >= 18 years old
* Receiving standard care (including antipsychotic and mood stabilizing medication)
* Mentally competent to give informed consent:

Exclusion Criteria:

* Substance use as cause of psychosis or (hypo)mania
* Substance use (other than nicotine) in the week prior to study onset
* Intellectual disability
* Diabetes mellitus (type 1 or type 2)
* Metabolic disease impacting ketone metabolism (NB: these are rare disorders diagnosed during childhood)
* Liver disease
* Kidney disease
* Cardiovascular disease
* Pregnancy
* Breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2024-12-01 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Prepulse Inhibition (PPI) - change dGK vs isocaloric control | measured 45 minutes (Tmax) after ingestion of intervention 1 (dGK) and 45 minuts after ingestion of intervention 2 (isocaloric carb control)
  PPI: an event-related potential (ERP) representing information processing (known to be disrupted in schizophrenia and bipolar disorder).
  The PPI task is an auditory paradigm featuring a total of 10 trials split evenly into two conditions: prepulse (PP) and non-prepulse (NP) in blocks. Startle pulses are 100dB at 40 ms, which is shown to provide significant startle visible in EEG126. Prepulse stimuli are 70 dB and 50 ms in duration, presented 50ms prior to the startle pulse. There is a 12 to 18 (avg: 15 s) interstimulus interval. All stimuli are white-noise blips. A calibrated apparatus is used to present the stimuli. Total estimated time is 20 min.

SECONDARY OUTCOMES:
P300 Event Related Potential (change dGK vs isocaloric control) | measured 65-75 minutes after ingestion of intervention 1 (dGK) and 75 minutes after ingestion of intervention 2 (isocaloric carb control); NB: directly after PPI.
  The P300 task consists of 160 stimuli in the oddball paradigm and requires the subjects to press a button on detection of the rare target (32/160). The common nontarget stimuli are 500 Hz, 100 ms duration. The rare target stimuli are 700 Hz. Both are 100 ms duration at 80 dB with variable interstimulus interval of 1.2 to 1.5 s. Preceded by 10 practice trials. This task has minimal burden and requires about 10 minutes.
Cognitive test: 15 Word Test (15WT) - change dGK vs isocaloric control | measured 75-85 minutes after ingestion of intervention 1 (dGK) and 75 minutes after ingestion of intervention 2 (isocaloric carb control); NB: directly after P300.
  15WT is a measure of verbal/episodic memory. The 15WT consists of 15 words, which have to be learned during three trials. After every trial the respondent is asked to recall as many words as possible. After a distraction period of 20 minutes, the respondent is asked to name the words they have learned before, again.
  Immediate recall after 1 test: maximum 15 words (minimum 0) Immediate recall after 3 test: maximum 45 words (minimum 0).
  Retention score after 20 minutes:
  1. percentage of correctly remembered words in the delayed recall-trial, relative to the number of words correctly remembered in the third immediate recall-trial
  2. percentage of correctly remembered words in the delayed recall-trial, relative to the maximum score in the immediate recall-trials
  Higher 15WT scores indicate better verbal/episodic memory, lower scores the opposite.
Cognitive test: Trail Making Test A (TMT-A) - change dGK vs isocaloric control | measured 75-85 minutes after ingestion of intervention 1 (dGK) and 75 minutes after ingestion of intervention 2 (isocaloric carb control); NB: directly after P300.
  TMT-A is a measure of (visual) attention. TMT-A outcome is the duration of time required to finalize test (including the time needed for the correction of errors prompted by the examiner), with a maximum of 5 minutes.
  The average TMT-A score in healthy adults is 29 seconds; a deficient score is greater than 78 seconds.
  Higher scores on TMT-A indicate worse (visual) attention.
Cognitive test: Trail-Making Test B (TMT-B) - (change dGK vs isocaloric control) | measured 75-85 minutes after ingestion of intervention 1 (dGK) and 75 minutes after ingestion of intervention 2 (isocaloric carb control); NB: directly after TMT-A.
  TMT-B is a measure of (frontal) executive functioning. TMT-B outcome is the duration of time required to finalize test (including the time needed for the correction of errors prompted by the examiner), with a maximum of 5 minutes.
  Average TMT-B score is 75 seconds; a deficient score is greater than 273 seconds.
  Higher scores on TMT-B indicate worse (frontal) executive functioning.
Cognitive test: Digit Span Test (DST) (change dGK vs isocaloric control) | measured 75-85 minutes after ingestion of intervention 1 (dGK) and 75 minutes after ingestion of intervention 2 (isocaloric carb control); NB: directly after TMT-B.
  DST is a measure for working memory. DST outcome is the maximum number of sequential digits correctly reproduced. In average healthy adults, the digit span is around 7 +/- 2. Minimum score is 0, maximum score is 9.
  Lower DST score indicate worse working memory.
Patient experience outcome on Mood, energy level, focus (change dGK vs isocaloric control) | measured circa 120 minutes after ingestion of intervention 1 (dGK) and circa 120 minutes after ingestion of intervention 2 (isocaloric carb control)
  visual analog scale (VAS) is used with a scale of 0 to 10 to measure patient-experiences effects of the interventions on their mood (0=extremely depression, 10 = extremely happy/euforic), energy level (0=completely exhauster, 10= extremely energetic) and ability to focus (0=completely unable to focus, 10=perfect focus).
Immune function: blood markers (change dGK vs isocaloric control) | first blood sample before ingestion (dGK or isocaloric control) (T0), then every 20 minutes in first hour after ingestion; afterwards every 30 minutes (max. 3 hours)
  sequential blood sampling through intravenous line: concentration (pg/ml) of inflammatory biomarkers relevant for immune function:
  * IL-1b
  * IL-6
  * IL-8
  * IL-10
  * TNF-a
  * IFN-g
  * hsCRP
  Comparison between dGK and isocaloric control at the same time points (see below).
Immune function: blood RNA markers (change dGK vs isocaloric control) | first blood sample before ingestion (dGK or isocaloric control) (T0), next at T0+90 minutes
  RNA expression analysis (immune panel nCounter, Nanostring) in whole blood: comparison dGK vs isocaloric control only at T0 plus 90 minutes.
Immune function: passive sweat IL-6 (change dGK vs isocaloric control) | Full 5 days of the study
  continuous measurement of IL-6 (pg/ml) in passive sweat (EnLiSense device)
Immune function: passive sweat TNF-a (change dGK vs isocaloric control) | Full 5 days of study
  continuous measurement of TNF-a (pg/ml)in passive sweat (EnLiSense device)
Metabolic function: Indirect Calorimetry (change dGK vs isocaloric control) | circa 90-120 minutes after ingestion of intervention 1 (dGK) and intervention 2 (isocaloric control); directly after finalizing cognitive tests.
  Resting energy expenditure (REE) is measured by gaseous exchange (indirect calorimetry). Oxygen consumption and CO2 production are measured during 20 minutes using a ventilated hood system (Q-NRG, Cosmed). Subjects lie flat on their backs and breathe into a canopy for 20 minutes. REE and Respiratory Quotient (RQ) are calculated with these measurements. The RQ represents the ratio of CO2 exhaled to the amount of 02 consumed by the individual and represents whole body substrate oxidation (glucose, fat and protein oxidation).
Metabolic function: blood biomarkers - change dGK vs isocaloric control | first blood sample before ingestion (both dGK and isocaloric control) (T0), then every 20 minutes in first hour after ingestion; afterwards every 30 minutes (max. 3 hours)
  Sequential blood sampling through intravenous line, to determine the plasma and serum concentrations of:
  * Glucose
  * Ketones
  * acylcarnitine profile
  * growth hormone (GH)
  * superoxide dismutase (SOD)
  * gluthione S-transferase (GST)
  * soluble intercellular adhesion molecule 1 (sICAM1)
  Comparison between dGK and isocaloric control at the same time points (see below).
Metabolic function: continuous glucose monitor (CGM) - change dGK vs isocaloric control | Full 5 days of the study.
  continuous glucose monitor (CGM; Abbott Libre Sense); continuous concentration in mM.
Circadian rhythm: passive sweat cortisol (change dGK vs isocaloric control) | Full 5 days of study
  continuous measurement of cortisol (pg/ml) in passive sweat (EnLiSense device)
Circadian rhythm: passive sweat melatonin (change dGK vs isocaloric control) | Full 5 days of study
  continuous measurement of melatonin (pg/ml) in passive sweat (EnLiSense device)

CONTACTS AND LOCATIONS:
Overall Officials: Karin Huizer, MD/PhD, Principal Investigator — Parnassia Groep
Locations (1):
- Amsterdam UMC, dept. Psychiatry, Amsterdam, North Holland, Netherlands

REFERENCES:
- [Derived] Dielemans DA, Yurtkap Y, van der Pluijm M, Soeters MR, Oranje B, Smit DJ, Ziermans T, van Tricht MJ, Muthukumar S, Prasad S, van der Mieden van Opmeer RL, Dekeyster E, Kamperman AM, Dyck JR, Rosema BS, Hoekstra R, Kupka RW, de Haan L, van Beveren NJ, Huizer K. The Effect of Exogenous Ketones on Signs and Symptoms of Schizophrenia Spectrum and Bipolar Disorders: Study Protocol for a Triple-Blind, Randomized, Controlled Crossover Pilot Study. Curr Dev Nutr. 2025 May 24;9(6):107480. doi: 10.1016/j.cdnut.2025.107480. eCollection 2025 Jun. PMID 40568354